CLINICAL TRIAL: NCT02741089
Title: Bronchoscopy Registry
Acronym: BSK
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Other Study IDs: 15-149
Record Dates: First submitted 2016-02-17; First posted 2016-04-18 (Estimated); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Indications for Flexible Bronchoscopy
Keywords: Analgosedation; Internal Quality Assurance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Serum, Blood plasm
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Indication for a flexible bronchoscopy: Patients representing to the hospital with the indication for a flexible bronchoscopy
  Interventions: Procedure: Indication for a flexible bronchoscopy

INTERVENTIONS:
Procedure: Indication for a flexible bronchoscopy — The data of patients are collected within the hospital routine documentation during the flexible bronchoscopy. The bronchoscopy is performed regardless of this study. Following the bronchoscopy the patients are asked a few questions about their health and their perception.
  The follow-up of all patients is done via phone calls in order to collect data about the outcome of each patient.

SUMMARY:
This monocentric, non-interventional observational registry study was designed in order to obtain data of patients with the indication for a flexible bronchoscopy to control and optimize a guideline conform therapy of these patients.

DETAILED DESCRIPTION:
Aims of this registry study are documentation of the characteristics of all patients with an indication for a flexible bronchoscopy who are attended at the University Hospital Aachen (UKA) to obtain new knowledge concerning safety and patient comfort using different medications for sedation.

Therefore a routine flexible bronchoscopy is carried out, whereat the choice of analgosedation medication is for the investigators decision, independent from the study.

Subsequently the following data are collected:

* duration of medical examination
* medication (e.g. midazolam, fentanyl, propofol, lidocain)
* vital signs at the end of the examination
* complications

Furthermore the patient should be asked concerning the general tolerance for the procedure and different symptoms like emesis, feeling of suffocation, cough and pain (0 = no stress, 100 = intolerable). In addition to that the grade of amnesia and the acceptance for later bronchoscopies should be asked.

Analyzing this data will optimize the internal quality control concerning the conducted examination, collect all complications related to the analgosedation and enhance the patients comfort during a flexible bronchoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Written declaration of consent
* Patients with the medical indication for a flexible bronchoscopy

Exclusion Criteria:

* Patients who are not fulfilling the inclusion criteria or:
* Pregnant or breastfeeding women
* Participation in other studies
* Sponsor-dependent patients or patients who are working with the sponsor
* Patients without mental ability or capacity to understand and follow the instructions of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with the medical indication for a flexible bronchoscopy by the attending physicians
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-02; Primary Completion 2020-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
demographic data | 20 minutes (before the routine intervention)
  Physiological parameters to assure internal quality control regarding the flexible bronchoscopy
indication for flexible bronchoscopy | 10 minutes (before the routine intervention)
  physiological parameters to assure internal quality control regarding the flexible bronchoscopy
smoking behaviour | 1 minute (before the routine intervention)
  physiological parameters to assure internal quality control regarding the flexible bronchoscopy
relevant side diseases | 10 minutes (before the routine intervention)
  physiological parameters to assure internal quality control regarding the flexible bronchoscopy
lung function parameters | 30 minutes (before the routine intervention)
  physiological parameters to assure internal quality control regarding the flexible bronchoscopy
anesthetic risk (ASA-Score) | 10 minutes (before the routine intervention)
  physiological parameters to assure internal quality control regarding the flexible bronchoscopy
vital signs | 10 minutes (before and after the routine intervention)
  physiological parameters to assure internal quality control regarding the flexible bronchoscopy
detection of complications depending on the different analgosedations | 30 minutes (during the routine intervention)
  physiological parameters to assure internal quality control regarding the flexible bronchoscopy
duration of medical examination | 30 minutes (during the routine intervention)
  physiological parameters to assure internal quality control regarding the flexible bronchoscopy
medication (e.g. midazolam, fentanyl, propofol, lidocain) | 5 minutes (after routine intervention)
  physiological parameters to assure internal quality control regarding the flexible bronchoscopy
general tolerance for the procedure and different symptoms like emesis, feeling of suffocation, cough and pain (0 = no stress, 100 = intolerable) | 5 minutes (after routine intervention)
  questionnaire
grade of amnesia | 5 minutes (after routine intervention)
  questionnaire
acceptance for later bronchoscopies | 5 minutes (after routine intervention)
  questionnaire

SECONDARY OUTCOMES:
identification of prognostic factors related to complications | 30 minutes (during the routine intervention)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dreher, Prof. Dr., Principal Investigator — RWTH Aachen University Hospital, MK1; Tobias Müller, PD, Principal Investigator — RWTH Aachen University Hospital, MK1
Locations (1):
- University Hospital Aachen, Department of Cardiology, Pneumology, Vascular Medicine and Intensive Care Medicine, Aachen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Undecided